CLINICAL TRIAL: NCT06803862
Title: RegiStry Of the multiFaceted medIcal cenTer
Acronym: SOFIT
Status: Active, not recruiting | Type: Observational
Sponsor: National Medical Research Center for Therapy and Preventive Medicine (Other Government)
Collaborators: State Healthcare Institution of the Tula Region Tula Regional Clinical Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: 01-10/22
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Chronic Non-communicable Diseases; Cardiovascular Diseases; COVID-19; Multimorbidity
Keywords: hospital registry; multifaceted medical center; cardiovascular diseases; multimorbidity; chronic non-communicable diseases
MeSH Terms: conditions — Noncommunicable Diseases; Cardiovascular Diseases; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a prospective medical registry (the SOFIT Registry) that enrolls all patients hospitalized in various departments of the Tula Regional Clinical Hospital in 2021.

The primary objective of the study is to analyze demographic, clinical and anamnestic characteristics of patients, history of COVID-19, the structure of multimorbidity, the quality of diagnostics and treatment, as well as short-term and long-term outcomes. As a part of this project a five-year follow-up is planned. The information will be obtained from Medical Information System resource of the hospital and regional and federal electronic databases.

DETAILED DESCRIPTION:
Nowadays in the Russian Federation chronic non-communicable diseases are one of the most common causes of hospitalization and also a concomitant pathology in the majority of patients undergoing hospital treatment in departments of various profiles. The creation of a prospective medical registry is an informative method for a comprehensive assessment of the characteristics of patients, including demographic, clinical and anamnestic data, the structure of multimorbidity, the quality of diagnostics and treatment as well as an assessment of short-term and long-term outcomes.

The aim of this project is to create a prospective registry of a multifaceted medical center (SOFIT), including all patients hospitalized in various departments of the hospital.

Patients admitted to the Tula Regional Clinical Hospital from 01.01.2021 to 31.12.2021 were retrospectively enrolled into this study. The information from electronic medical records was obtained using the Medical Information System resource of the hospital.

At the first stage, it is planned to analyze the age and gender characteristics of patients, the proportion of cases of cardiovascular and chronic non-cardiac diseases and their combinations, the frequency of a history of COVID-19, laboratory and instrumental data, cardiovascular pharmacotherapy prescribed in the hospital and hospital mortality. The obtained data will be compared in the cardiologic, therapeutic and other departments.

At the second stage, the prospective follow-up will be carried out up to 5 years after the reference hospitalization. It will involve the evaluation of long-term outcomes, such as all-cause mortality, cardiovascular events (cardiovascular death, nonfatal myocardial infarction, nonfatal cerebral stroke, hospitalizations and surgical interventions for cardiovascular diseases), cases of COVID-19 based on patient's medical records. The information about cases of death (date and cause of death, place of death registration), cardiovascular events during follow-up will be obtained from the regional database of death cases in population of the Tula region and from other regional electronic databases. The information about cases of COVID-19 will be obtained from the Russian Federal Registry of COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. Patients hospitalized to the Tula Regional Clinical Hospital from 01.01.2021 to 31.12.2021.
2. Age 18 years and older.
3. Permanent residency in Tula city and Tula region.

Exclusion Criteria:

1. Permanent residency outside of Tula city and Tula region.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the Tula Regional Clinical Hospital from 01.01.2021 to 31.12.2021 who meet inclusion criteria and don't have exclusion criteria will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 21783 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 5 years after inclusion
Time to all-cause mortality, cardiovascular mortality, nonfatal myocardial infarction, nonfatal cerebral stroke, coronary/carotid revascularization | from discharge up to 5 years after reference hospitalization

SECONDARY OUTCOMES:
Time to composite endpoint (nonfatal myocardial infarction or nonfatal cerebral stroke or coronary/carotid revascularization) | from discharge up to 5 years after reference hospitalization
Proportion of patients with nonfatal myocardial infarction | from discharge up to 5 years after reference hospitalization
Proportion of patients with nonfatal cerebral stroke | from discharge up to 5 years after reference hospitalization
Proportion of patients with cases of COVID-19 during follow-up | from discharge up to 5 years after reference hospitalization
Hospitalization due to cardiovascular disease, proportion of patients with hospitalization due to cardiovascular disease | from discharge up to 5 years after reference hospitalization
Hospitalization due to COVID-19, proportion of patients with hospitalization due to COVID-19 | from discharge up to 5 years after reference hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail M Loukianov, MD, PhD, Study Chair — National Medical Research Center for Therapy and Preventive Medicine; Tatyana A Gomova, MD, PhD, Study Chair — State Healthcare Institution of the Tula Region Tula Regional Clinical Hospital; Ruslan N Shepel, MD, PhD, Study Chair — National Medical Research Center for Therapy and Preventive Medicine; Oxana M Drapkina, MD, PhD, professor, Study Chair — National Medical Research Center for Therapy and Preventive Medicine
Locations (2):
- Russia (2):
  - National Research Center for Preventive Medicine of the Ministry of Health, Moscow
  - State Healthcare Institution of the Tula Region Tula Regional Clinical Hospital, Tula

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ignatieva VI, Kontsevaya AV, Lukyanov MM, et al. Cost-effectiveness analysis of increasing drug therapy coverage for patients with coronary artery disease in combination with atrial fibrillation and heart failure. Cardiovascular Therapy and Prevention. 2024;23(4):3950. (In Russ.) https://doi.org/10.15829/1728-8800-2024-3950
- [Result] Loukianov MM, Gomova TA, Savishceva AA, et al. RegiStry Of the multiFaceted medIcal cenTer (SOFIT): the main tasks, development, and the first results. Russian Journal of Preventive Medicine. 2023;26(6):46 54. (In Russ.) https://doi.org/10.17116/profmed20232606146